CLINICAL TRIAL: NCT03446547
Title: Ablative STEreotactic RadiOtherapy wIth Durvalumab (MEDI4736). An Open Label Randomized Phase II Trial With Durvalumab Following Stereotactic Body Radiotherapy (SBRT) in Patients With Stage I Non-small Cell Lung Cancer (NSCLC)
Brief Title: Ablative STEreotactic RadiOtherapy wIth Durvalumab (MEDI4736)
Acronym: ASTEROID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Andreas Hallqvist, Principal Investigator, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-005225-37
Record Dates: First submitted 2018-02-11; First posted 2018-02-27 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: NSCLC, Stage I
Keywords: SBRT; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (No Intervention): SBRT and follow-up
- Arm B (Experimental): SBRT followed by Durvalumab
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — durvalumab 1500 mg i.v. every fourth week for 12 months
  Other Names: Medi4736
  Arms: Arm B

SUMMARY:
This is a randomized multicentre open label phase II study of Durvalumab following Stereotactic Body Radiotherapy (SBRT) in patients with T1-2N0M0 NSCLC.

Patients will be randomized 1:1 to follow up or receiving Durvalumab every 4th week for 12 months

DETAILED DESCRIPTION:
This is a randomized multicentre open label phase II study of the PDL1 inhibitor Durvalumab following SBRT in patients with T1-2N0M0 NSCLC. It will enroll 106 patients aiming at a minimum of 5 subjects per site. The subjects will be randomized in a 1:1 fashion with performance status, gender and T-stage as stratification factors. Patients with peripheral lung tumors will receive SBRT usually between 3 and 4 fractions. The group randomized to immunotherapy will then receive Durvalumab, given with a fixed dose of 1500 mg i.v. every fourth week during 12 months. Both arms will be assessed according to the same follow-up schedule with radiology every third month.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to performing any protocol- related procedures, including screening evaluations
* Histological or cytological diagnosis of NSCLC
* Stage I-IIA tumours ≤ 5 cm
* Peripheral tumours
* Medically inoperable patients or patients refusing surgery
* Received no prior chemotherapy or radiation therapy for NSCLC
* Age > 18 years at time of study entry, no upper age limit
* WHO performance status 0-2
* Adequate normal organ and marrow function as defined below:
* Haemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
* Platelet count ≥ 100 x 109/L (>100,000 per mm3)
* Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* AST/ALT ≤ 2.5 x institutional upper limit of normal
* Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by chrome-EDTA or Iohexol clearance
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Centrally located tumours
* No regional or distant metastases are allowed (i.e. no stage II-IV disease)
* Oxygen usage or a FEV1 < 0.7 L and CO diffusion capacity < 30%
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 4 weeks
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
* Second primary residual malignancy. Other malignancy diagnosed and treated > 5 years ago without relapse is allowed. (Carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin < 5 years are allowed)
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Active or prior documented autoimmune or inflammatory disorders . The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Subjects without active disease in the last 5 years may be included but only after consultation with the study physician
  * Subjects with celiac disease controlled by diet alone
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NYHA III-IV), uncontrolled hypertension, unstable angina pectoris, interstitial lung disease, cardiac arrhythmia, active peptic ulcer disease, active bleeding diatheses
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
* Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
TTP | From date of randomization until the date of first documented progression, assessed up to 60 months
  Time to progression

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 60 months
  Overall survival
LC | Assessed at scheduled timepoints every 3-6 months through study completion (60 months)
  Local control
QoL | Measured at baseline and at three timepoints (6, 12 and 20 months)
  QoL by LCSS
TTP by PDL1 expression | From date of randomization until the date of first documented progression, assessed up to 60 months
  Time to progression related to level of PDL1expression

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hallqvist, PhD, Principal Investigator — Göteborg University
Locations (15):
- Finland (4):
  - Helsinki, Helsinki
  - Dept of Oncology, Tampere
  - Turku, Turku
  - Dept of Oncology, Vaasa
- Norway (4):
  - Ålesund, Ålesund
  - Dept of Oncology, Oslo
  - Dept of pulmonary medicine, Tromsø
  - Dept of Oncology, Trondheim
- Sweden (7):
  - Dept of pulmonary medicine, Gävle
  - Dept. of Oncology, Gothenburg
  - Dept of pulmonary medicine, Linköping
  - Sunderbyn, Luleå
  - Dept of pulmonary medicine, Lund
  - Dept of Oncology, Stockholm
  - Dept. of Oncology, Umeå

IPD SHARING:
Plan to Share IPD: No
Will be available later on